CLINICAL TRIAL: NCT07190755
Title: Impact of Patient-Reported Outcomes for Symptom Monitoring in Patients Followed for Curative Treatment of Head and Neck Squamous Cell Carcinoma (HNSCC) With Radiotherapy or Chemoradiotherapy
Brief Title: Impact of Patient-Reported Outcomes for Symptom Monitoring in Patients Followed for Head and Neck Squamous Cell Carcinoma (HNSCC)
Acronym: WEBNECK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Collaborators: Resilience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHB24.06
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma HNSCC
Keywords: head and neck squamous cell carcinoma; symptoms monitoring; web monitoring
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (No Intervention): patients will be followed as standard of care
- remote symptoms monitoring (Experimental): Participants in the intervention arm will use Resilience PRO, a mobile phone application regularly asking participants about their symptoms. For clinically important symptoms, an alert is sent to the care team that can incorporate that information to timely adjust the care of the participants.
  Interventions: Other: Remote symptoms moniotring

INTERVENTIONS:
Other: Remote symptoms moniotring — Participants in the intervention arm will use Resilience PRO, a mobile phone application regularly asking participants about their symptoms. For clinically important symptoms, an alert is sent to the care team that can incorporate that information to timely adjust the care of the participants.
  Arms: remote symptoms monitoring

SUMMARY:
The use of digital strategies to systematically monitor patients' symptoms in clinical settings allows problems to be detected at an early stage before they worsen or lead to complications. In this study, the hypothesis is that the proportion of patients with a weight loss of at least 5% between before radiotherapy/radiochemotherapy and 3 months after treatment would be lower with optimised care thanks to remote monitoring using a medical telemonitoring solution in oncology.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 and under 75 years WHO score < 2,

  * Treated for localised heand and neck cancer of the squamous cell carcinoma type for which curative treatment has been chosen and receiving radiotherapy or radio-chemotherapy exclusively or as an adjuvant with the aim of cure
  * Having signed the informed consent form,
  * Affiliated with or beneficiary of a social protection scheme,
  * Access to a smartphone or the internet,

Exclusion Criteria:

* History of other neoplastic disease less than 2 years ago or progressive disease,
* History of ENT radiotherapy,
* Pregnant or breastfeeding women,
* Protected adults (under guardianship, curatorship or judicial protection),
* Patients participating in a therapeutic study,
* Patients unable to understand the study for any reason or to comply with the constraints of the trial (language, psychological or geographical issues, etc.), patients with blindness preventing the use of the medical telemonitoring solution in oncology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Impact of remote monitoring of symptoms on weight loss | 3 months after treatment
  Proportion of patients with at least a 5% reduction in weight 3 months after treatment compared to the consultation at the start of radiotherapy or radiochemotherapy

SECONDARY OUTCOMES:
Impact of remote symptoms monitoring on global survival | 12 month after treatment
  Time beetween inclusion and death for any cause
Impact of remote symptoms monitoring on global survival | 18 month after treatment
  Time beetween inclusion and death for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Thureau, MD,PhD, Principal Investigator — Centre Henri Becquerel
Locations (2):
- France (2):
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No